CLINICAL TRIAL: NCT00333281
Title: A Randomized, Double-Blind, Parallel-Design, Placebo-Controlled Study to Evaluate the Effects of 5 mg Tadalafil (IC351, LY450190) and 50 mg Sildenafil Administered Once Daily for 6 Months on Visual Function in Healthy Subjects or Subjects With Mild Erectile Dysfunction
Brief Title: A Study of Visual Effects of Erectile Dysfunction Medications Dosed Daily for Six Months
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9520; H6D-MC-LVGO
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Erectile Dysfunction
Keywords: Healthy Volunteers
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

INTERVENTIONS:
Drug: tadalafil
  Other Names: LY450190; Cialis; IC351

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the effects on vision of six months of daily dosing of 5 mg tadalafil or 50 mg sildenafil compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or males with mild erectile dysfunction (ED).
* Between the ages of 30 and 65 years, inclusive.

Exclusion Criteria:

* Phosphodiesterase type 5 (PDE5) inhibitor therapy (tadalafil, sildenafil, or vardenafil) within 6 weeks of the start of the study.
* Diagnosis of diabetes mellitus.
* Any chronic illness or medication that is a risk factor for eye disease or any medication that causes retinal toxicity or affects visual function.
* Certain chronic medical conditions including unstable angina pectoris, severe renal [kidney] insufficiency, clinically significant hepatobiliary [liver, bile duct] disease, cancer, and AIDS/HIV.
* A history of clinically significant chronic ophthalmologic disease or any significant visual abnormality identified at the start of the study.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198
Dates: Start 2005-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in dark-adapted bright flash b-wave amplitude on electroretinography (ERG) testing at baseline, 3 & 6 months on drug, and 4-6 weeks after discontinuation of drug.

SECONDARY OUTCOMES:
Five other ERG waveform components; intraocular pressure; visual acuity; peripheral vision; color discrimination; and inspection of anterior chamber, lens, and retinal anatomy.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Cordell WH, Maturi RK, Costigan TM, Marmor MF, Weleber RG, Coupland SG, Danis RP, McGettigan JW Jr, Antoszyk AN, Klise S, Sides GD; ERG Testing During Chronic PDE5 Inhibitor Administration (ERG-PDE5i) Consortium. Retinal effects of 6 months of daily use of tadalafil or sildenafil. Arch Ophthalmol. 2009 Apr;127(4):367-73. doi: 10.1001/archophthalmol.2009.36. PMID 19365010
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com